CLINICAL TRIAL: NCT06186921
Title: Effect of Different Intraligamentary Injections on the Post-endodontic Pain in Patients With Symptomatic Irreversible Pulpitis
Brief Title: Intraligamentary Injections and Post-endodontic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jamia Millia Islamia (Other)
Responsible Party: Principal Investigator, Dr. Vivek Aggarwal, Professor, Jamia Millia Islamia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Postendo pain Intraligamentary
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Pulpitis
MeSH Terms: conditions — Pulpitis | interventions — Dexamethasone; Diclofenac; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intraligamentary injection of dexamethasone (Experimental): After endodontic instrumentation and placement of temporary restoration, the patients shall receive Intraligamentary injection of dexamethasone
  Interventions: Drug: Dexamethasone
- Intraligamentary injection of diclofenac sodium (Experimental): After endodontic instrumentation and placement of temporary restoration, the patients shall receive Intraligamentary injection of dexamethasone
  Interventions: Drug: Dexamethasone
- Intraligamentary injection of 0.5% bupivacaine (Experimental): After endodontic instrumentation and placement of temporary restoration, the patients shall receive Intraligamentary injection of dexamethasone
  Interventions: Drug: Dexamethasone
- Intraligamentary injection of 2% lidocaine (Active Comparator): After endodontic instrumentation and placement of temporary restoration, the patients shall receive Intraligamentary injection of dexamethasone
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — After endodontic instrumentation and placement of temporary restoration, the patients shall receive intraligamentary injections.
  Other Names: diclofenac sodium; bupivacaine

SUMMARY:
This study will aim to evaluate postoperative pain after intraligamentary injections of dexamethasone (4mg/ml), diclofenac sodium (25mg/ml), 0.5% bupivacaine and 2% lidocaine given to the patients with symptomatic irreversible pulpitis after completion of the first appointment. Objectives: 1. To evaluate postoperative pain in patients receiving intraligamentary injections of either dexamethasone (4mg/ml), diclofenac sodium (25mg/ml), 0.5% bupivacaine or 2% lidocaine. 2. To compare the postoperative pain in different groups.

DETAILED DESCRIPTION:
The patients will receive a primary Inferior alveolar nerve block injection using 1.8 mL of 2% lidocaine with 1: 80 000 epinephrine using a direct Halsted approach. The needle will be inserted until bony resistance is felt. After reaching the target area, aspiration will be performed, and the solution will be deposited over 60 seconds. After 10 minutes, the patients will be asked about the lip numbness. Patients without profound lip numbness will be excluded from the study since the block will be considered as 'missed'. A conventional access opening will be initiated after isolation with a rubber dam. After endodontic instrumentation and placement of temporary restoration, the patients shall receive intraligamentary injections of dexamethasone (4mg/ml), diclofenac sodium (25mg/ml), 0.5% bupivacaine, and 2% lidocaine. The patients will be randomly allocated to treatment groups with the help of an online random generator. The presence of postoperative pain (using Heft Parker visual analog pain scale) will be assessed at 2 hours, 6 hours, 24 hours, and 72 hours after treatment. The pain score proforma shall be collected at the subsequent visit.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic carious exposed mandibular first or second molars.
* Positive and prolonged response to thermal sensitivity tests and electric pulp tests.
* Vital coronal pulp on access cavity preparation.
* American Society of Anesthesiologists class I or II medical history.
* Ability to understand the use of pain scales.

Exclusion Criteria:

* Active pain in more than 1 tooth
* Teeth with fused roots.
* Radiographic evidence of an extra root.
* Large restorations with overhanging margins.
* Full crowns or deep periodontal pockets.
* Known allergy or contraindications to any content of the local anesthetic solution or NSAIDs
* History of known or suspected drug abuse.
* Taking any drugs which could affect the pain perception, e.g, opioids, antidepressants, anticonvulsants, muscle relaxants, anxiolytics, sedatives, NSAIDs.
* Pregnant or breastfeeding patients.
* Patients with asthma, gastric ulcers, and bleeding disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-12-02 (Actual); Primary Completion 2024-03-03 (Estimated); Study Completion 2024-03-03 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 2 hours, 6 hours, 24 hours and 72 hours after treatment
  The presence of postoperative pain (using Heft Parker visual analog pain scale) will be assessed at 2 hours, 6 hours, 24 hours and 72 hours after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Jamia MIliia Islamia, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes